CLINICAL TRIAL: NCT04229589
Title: Risk of Syncopal Relapses in Patients Treated With Permanent Pacing for Bradyarrhythmic Syncope
Acronym: SYNCOPACED
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Sponsor
Other Study IDs: SYNCOPACED
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Syncope
Keywords: Syncope, pacemaker, bradyarrhythmias
MeSH Terms: conditions — Syncope; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Consecutive patients undergoing pacemaker implantation for bradyarrhythmic syncope
  Interventions: Other: Clinic follow-up

INTERVENTIONS:
Other: Clinic follow-up — Patients are regularly evaluated to asses the occurrence of syncopal relapses

SUMMARY:
Prospective, multicenter, observational registry designed to collect data on syncopal relapses in patients undergoing pacemaker implantation for bradyarrhythmic syncope.

DETAILED DESCRIPTION:
Prospective, multicenter, observational registry designed to collect data on syncopal relapses in patients undergoing pacemaker implantation for bradyarrhythmic syncope. All consecutive patients aged ≥18 years who underwent pacemaker implantation for syncope of bradyarrhythmic aetiology (proven or presumed) at participating centers from January 2010 to December 2013 were enrolled in the registry. During follow-up the occurrence of the first syncopal relapse after pacemaker implantation is recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing pacemaker implantation for bradyarrhythmic syncope

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing pacemaker implantation for bradyarrhythmic syncope (proven or presumed) according current guidelines
Sampling Method: Non-Probability Sample
Enrollment: 1364 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Syncopal relapse | march 2020
  First syncopal relapse after pacemaker implantation

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - "Card. G. Panico" Hospital, Tricase, Lecce
  - Federico Guerra, Ancona
  - Policlinico S.Orsola-Malpighi, Bologna
  - AO Pugliese-Ciaccio, Catanzaro
  - Monaldi Hospital, Napoli
  - AOU "Maggiore della Carità", Novara
  - Dell'Era Gabriele, Novara

IPD SHARING:
Plan to Share IPD: No